CLINICAL TRIAL: NCT00684658
Title: An Internet Coping Skills Training Program for Teens With Type 1 Diabetes
Brief Title: TEENCOPE: An Internet Coping Skills Training Program for Teens With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0711003291; R01NR004009 (NIH)
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Children and Teenagers; Coping with Chronic Illness; Adolescence; Internet psychosocial program; Coping Skills Training
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): TeenCope: Internet-based Coping Skills Training
  Interventions: Behavioral: TeenCope
- 2 (Active Comparator): Managing Diabetes: Internet-based Diabetes Education
  Interventions: Behavioral: Managing Diabetes

INTERVENTIONS:
Behavioral: TeenCope — Teencope consists of a series of 5 sessions designed to increase children's sense of competence and mastery by retraining inappropriate or non-constructive coping styles and forming more positive styles and patterns of behavior. Each week a new 30-45 minute session is uploaded to a password-protected website on the Yale server for youth to complete. Youth are grouped with 8-12 peers who complete the same weekly sessions in an asynchronous manner. Youth interact with each other on an online discussion board moderated by a clinical psychologist
  Arms: 1
Behavioral: Managing Diabetes — Managing Diabetes consists of 5 sessions on educational content related to diabetes self management targeted to adolescents. As with the TeenCope program, each week a new 30-45 minute session is uploaded to a password-protected website on the Yale server for youth to complete. Youth complete educational sessions independently over 5 weeks. There is no online discussion board or peer interaction.
  Arms: 2

SUMMARY:
The purpose of the study is to compare the effects of a 5-week internet-based coping skills training program (TeenCope) with a 5-week internet education program (Managing Diabetes) in youth (age 11-14) with type 1 diabetes on intensive insulin therapy.

DETAILED DESCRIPTION:
It is well established that for many youth with type 1 diabetes (T1D), the developmental stage of puberty is characterized by a significant deterioration in metabolic control. Previous research conducted by the Yale School of Nursing demonstrates that providing cognitive-behavioral coping skills training program (CST) as a supplement to intensive medical treatment regimen enhances physiological and psychosocial outcomes - most notably in youth as they approach adolescence. Successful CST programs studied at Yale consist of weekly, in-person group sessions over a 5-week period conducted by a clinical psychologist or social worker.

Rapid advances in technology have made the internet a compelling tool to reach out to youth and significantly broaden the application of CST programs. Investigators at Yale (scientists, NPs, clinical psychologists) have teamed with web specialists (computer programmers, web designers, graphic artists, and illustrators) and youth with T1D and their parents to adapt the successful CST program for use on the internet. In this trial, internet-based CST (TeenCope) will be evaluated by comparing it to an internet-based education program for managing diabetes (Managing Diabetes).

Three hundred (300) youth from 4 different sites within the U.S will take part in the study. Youth will be randomly assigned to complete either the TeenCope or Managing Diabetes program right away, and will be given the opportunity to complete the alternate program after 12 months. Data on psychosocial and disease management parameters will be collected at baseline, 3, 6, 12 and 18 months through youth filling out online questionnaires (lasting approximately 30 minutes). Clinical outcome data (height, weight, HbA1c, episodes of hypoglycemia, DKA, and hospitalization) will be collected from the medical chart throughout the study, and parents will complete a demographic data form.

This study has great potential for working with youth with type 1 diabetes. If proven effective, the investigators are interested in continued dissemination and translation of this intervention beyond their geographical location.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-14
* English speaking
* Youth assents and parent consents to participation
* School grade is appropriate to age within 1 year
* Type 1 diabetes for a minimum of 6 months
* Access to high speed internet service for 5 week intervention (will be arranged by study if not presently in the home)

Exclusion Criteria:

* Other significant chronic health problems requiring intensive self-management
* Previous exposure to Yale School of Nursing's Coping Skills Training or Managing Diabetes materials

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | 18 months
Pediatric Quality of Life Inventory (PedsQL) | 18 months

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | 18 months
Self-Efficacy for Diabetes Scale | 18 months
Children's Depression Inventory | 18 months
Self-Perception Profile for Adolescents | 18 months
Responses to Stress Questionaire (RSQ) | 18 months
Diabetes Family Behavior Scale | 18 months
Self Management of Type 1 Diabetes | 18 months
Diabetes Conflict | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Grey, DrPh, FAAN, CPNP, Principal Investigator — Yale School of Nursing; Robin Whittemore, PhD, APRN, Principal Investigator — Yale School of Nursing
Locations (4):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - Yale University School of Nursing, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Grey M, Boland EA, Davidson M, Li J, Tamborlane WV. Coping skills training for youth with diabetes mellitus has long-lasting effects on metabolic control and quality of life. J Pediatr. 2000 Jul;137(1):107-13. doi: 10.1067/mpd.2000.106568. PMID 10891831
- [Background] Grey M, Boland EA, Davidson M, Yu C, Sullivan-Bolyai S, Tamborlane WV. Short-term effects of coping skills training as adjunct to intensive therapy in adolescents. Diabetes Care. 1998 Jun;21(6):902-8. doi: 10.2337/diacare.21.6.902. PMID 9614605
- [Background] Whittemore R, Grey M, Lindemann E, Ambrosino J, Jaser S. Development of an Internet coping skills training program for teenagers with type 1 diabetes. Comput Inform Nurs. 2010 Mar-Apr;28(2):103-11. doi: 10.1097/NCN.0b013e3181cd8199. PMID 20182161
- [Background] Grey M, Whittemore R, Liberti L, Delamater A, Murphy K, Faulkner MS. A comparison of two internet programs for adolescents with type 1 diabetes: design and methods. Contemp Clin Trials. 2012 Jul;33(4):769-76. doi: 10.1016/j.cct.2012.03.012. Epub 2012 Mar 29. PMID 22484337
- [Derived] Jaser SS, Whittemore R, Chao A, Jeon S, Faulkner MS, Grey M. Mediators of 12-month outcomes of two Internet interventions for youth with type 1 diabetes. J Pediatr Psychol. 2014 Apr;39(3):306-15. doi: 10.1093/jpepsy/jst081. Epub 2013 Oct 26. PMID 24163439
- [Derived] Grey M, Whittemore R, Jeon S, Murphy K, Faulkner MS, Delamater A; TeenCope Study Group. Internet psycho-education programs improve outcomes in youth with type 1 diabetes. Diabetes Care. 2013 Sep;36(9):2475-82. doi: 10.2337/dc12-2199. Epub 2013 Apr 11. PMID 23579179
- [Derived] Whittemore R, Jaser SS, Jeon S, Liberti L, Delamater A, Murphy K, Faulkner MS, Grey M. An internet coping skills training program for youth with type 1 diabetes: six-month outcomes. Nurs Res. 2012 Nov-Dec;61(6):395-404. doi: 10.1097/NNR.0b013e3182690a29. PMID 22960587
- [Derived] Jaser SS, Faulkner MS, Whittemore R, Jeon S, Murphy K, Delamater A, Grey M. Coping, self-management, and adaptation in adolescents with type 1 diabetes. Ann Behav Med. 2012 Jun;43(3):311-9. doi: 10.1007/s12160-012-9343-z. PMID 22274724